CLINICAL TRIAL: NCT05786963
Title: Comparison of Hepatus and FibroScan for Evaluation of Fibrosis and Steatosis in Chronic Hepatitis B or NAFLD Patients
Brief Title: Comparison of Hepatus and FibroScan for Evaluation of Fibrosis and Steatosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hong You, Vice President of Beijing Friendship Hospital, Beijing Friendship Hospital
Other Study IDs: YYYXYJ-2022-095
Record Dates: First submitted 2022-11-27; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Chronic Hepatitis b; Non-Alcoholic Fatty Liver Disease
Keywords: Chronic Hepatitis b; Non-alcoholic Fatty Liver Disease; Liver fibrosis/cirrhosis; Steatosis
MeSH Terms: conditions — Hepatitis B, Chronic; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Fibrosis; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Totals of 400 chronic hepatitis B or non-alcoholic fatty liver disease (NAFLD) patients with or without cirrhosis will be enrolled. Patients' clinical characteristics, including alanine aminotransferase, aspartic aminotransferase, total bilirubin, direct bilirubin, indirect bilirubin, triglyceride and total cholesterol, hepatitis B surface antigen, steatosis, and liver stiffness measurement will be collected. The consistence of liver fibrosis and steatosis assessment between Hepatus and FibroScan will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with or without cirrhosis diagnose as chronic hepatitis B or non-alcoholic fatty liver disease;
* Age above 18 years;
* Signature of informed consent.

Exclusion Criteria:

* Patients with HCV and/or other viral hepatitis, autoimmune liver disease, alcoholic liver disease, genetic liver disease or other chronic liver diseases;
* Patients with decompensated cirrhosis;
* Patients with serum total bilirubin level higher than 51 umol/L;
* Patients with liver malignant lesion, hemangiomas, giant liver cysts and other liver lesions;
* Patients with HIV infections;
* Patients after liver transplantation or TIPS;
* Pregnant women;
* Patients with Budd-Chiari syndrome, chronic congestive heart failure, constrictive pericarditis or other liver congestion lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without cirrhosis diagnose as chronic hepatitis B or non-alcoholic fatty liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Consistency of liver stiffness and steatosis results in the same location between Hepatus in continuous measurement mode and FibroScan in single detection mode. | 1 to 3 years
  Consistency of liver stiffness and steatosis between Hepatus and FibroScan.

SECONDARY OUTCOMES:
Consistency of liver stiffness and steatosis results between Hepatus in continuous measurement mode and FibroScan in single detection mode through the respective localization methods. | 1 to 3 years
  The localization method of Hepatus is the real-time two-dimensional image guiding system, which is manually location in FibroScan.
Consistency of liver stiffness and steatosis results between Hepatus and FibroScan in single detection mode. | 1 to 3 years
  The localization methods include the respective localization methods in Hepatus and FibroScan, and manually locating.
Comparison of measurement performance in Hepatus under continuous detection mode and in FibroScan through single detection mode. | 1 to 3 years
  Evaluation of measurement performance includes the rate of successful detection, time taken for validated detection, stability of liver stiffness measurement and controlled attenuation parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Hong You, doctor, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Yameng Sun, Beijing, Select A State Or Province, China